CLINICAL TRIAL: NCT00732199
Title: Determinants of Age-specific Breathing Instability During Sleep
Brief Title: Determinants of Age Related Breathing Instability During Non-Rapid-Eye-Movement (NREM) Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CDA-2-019-07F
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-04

CONDITIONS: Sleep Apnea; Age
Keywords: apneic threshold; central apnea; intermittent hypoxia; aging; ventilation; chemoresponsiveness; carbon-dioxide reserve
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Central; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Other): Determine the apneic threshold and carbon- dioxide reserve using noninvasive positive pressure ventilation during NREM sleep and determine the effect effect of episodic hypoxia on ventilatory long-term facilitation during NREM sleep in Young adults.
  Interventions: Other: 1) hyperventilation via noninvasive positive pressure ventilation 2) multiple trials of episodic hypoxia
- Arm 2 (Experimental): Determine the apneic threshold and carbon- dioxide reserve using noninvasive positive pressure ventilation during NREM sleep and determine the effect of episodic hypoxia on ventilatory long-term facilitation during NREM sleep in Older adults.
  Interventions: Other: 1) hyperventilation via noninvasive positive pressure ventilation 2) multiple trials of episodic hypoxia

INTERVENTIONS:
Other: 1) hyperventilation via noninvasive positive pressure ventilation 2) multiple trials of episodic hypoxia — 1) noninvasive hyperventilation to determine apneic threshold; 2) episodic hypoxia to determine ventilatory long term facilitation

SUMMARY:
The purpose for this research protocol was to examine the role of breathing control mechanisms that determine the development of sleep-disordered breathing in the elderly. This proposal focused on key factors that contribute to the control of ventilation in elderly adults during sleep. The investigators studied the age-specific changes in ventilatory control in older and young adults during NREM sleep.

DETAILED DESCRIPTION:
Sleep apnea-hypopnea syndrome (SAS) is a relatively common disorder in the US population with significant adverse health consequences. Despite the high prevalence of SAS in elderly individuals, the underlying mechanisms have remained elusive. Specifically, the investigators do not know whether the high prevalence of sleep apnea in older adults is due to increased central breathing instability. This proposal focused on investigating age-specific differences in the susceptibility to central breathing instability in adults.

This project had the following specific objectives:

* To determine age-specific changes in the hypocapnic apneic threshold during NREM sleep in elderly vs young individuals.
* To determine age-specific changes in long-term facilitation during sleep in elderly versus young individuals.

Procedure: The investigators determined the susceptibility to central breathing instability by mechanically ventilating the subjects during NREM sleep using non-invasive pressure support ventilation. The investigators compared the hypocapnic apneic threshold in old (age>60 years) and young (age 18-50 years) individuals who were healthy. The investigators also measured the parameters over a continuum of age from 18 to 89 years.

- The investigators investigated whether there was a difference in the susceptibility to long term facilitation of ventilation between young and old healthy individuals in response to episodic hypoxia, while maintaining isocapnia.

Sleep apnea is very common in older Veterans and is associated with significant cardiovascular complications. Greater insight into the pathogenesis will have a positive impact on the health of Veterans suffering from this condition. This study furthers the understanding of the pathogenesis of breathing instability leading to sleep-disordered breathing during sleep. The investigators anticipate findings will provide a basis for new approaches to prevention and management of SAS in Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy older and young adults

Exclusion Criteria:

* Pregnancy,
* history of active coronary artery disease-including stable and unstable angina,
* recent myocardial infarction,
* history of congestive heart failure,
* stroke,
* excessive daytime sleepiness with Epworth Sleepiness Scale of >15
* patient with OSA- (Obstructive sleep apnea) on therapy
* depression,
* schizophrenia,
* untreated hypothyroidism,
* diabetes on insulin,
* seizure disorder,
* intrinsic renal and liver disorders,
* failure to give informed consent,
* patients with evidence of pulmonary diseases based on history and abnormal pulmonary function testing, including obstructive (ratio of predicted forced expiratory volume to forced vital capacity, <80% predicted) or restrictive lung disorders (total lung capacity <80% predicted) with resting oxygen saturation of <96% and kyphoscoliosis (chest wall deformities)
* patients on certain medications including, opiates derivatives, stimulants, antidepressants, tranquilizers, anti-psychotic agents, theophylline and other central nervous system altering medications
* history of alcohol or recreational drug use will also serve as grounds for exclusion,
* patients with body mass index (BMI) >34kg/m2
* subjects with sleep apnea are already using continuous positive airway pressure for more than 7 days as therapy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2008-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susmita Chowdhuri, MD, Principal Investigator — John D. Dingell VA Medical Center, Detroit, MI
Locations (1):
- John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chowdhuri S, Pranathiageswaran S, Franco-Elizondo R, Jayakar A, Hosni A, Nair A, Badr MS. Effect of age on long-term facilitation and chemosensitivity during NREM sleep. J Appl Physiol (1985). 2015 Nov 15;119(10):1088-96. doi: 10.1152/japplphysiol.00030.2015. Epub 2015 Aug 27. PMID 26316510

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by posting fliers at the sites approved by the Detroit VA clinical investigations committee and Wayne State IRB (institution review board). They completed a phone interview. If they qualified based on the inclusion/exclusion criteria they completed an informed consent. Dates 2008 to 2014.
Groups:
- Arm 1: Young adults, age 18-59yrs
  hyperventilation and episodic hypoxia: a) noninvasive hyperventilation to determine apneic threshold; b) episodic hypoxia to determine ventilatory long term facilitation
- Arm 2: Older adults, age >/=60 yrs
  hyperventilation and episodic hypoxia: a) noninvasive hyperventilation to determine apneic threshold; b) episodic hypoxia to determine ventilatory long term facilitation
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 50 | 42
Completed | 16 | 16
Not Completed | 34 | 26
Not completed — Withdrawal by Subject | 25 | 18
Not completed — sleep apnea, inadequate signals/sleep | 9 | 8

BASELINE CHARACTERISTICS:
Population: We studied normal subjects. Subjects were assigned to two age categories, 'young' between 18 and 50 years, and 'elderly' >55-60 years respectively. Participants with data available were included in the analysis Normal participants (controls) will have apnea hypopnea index, AHI<5/hour, respiratory events /hour of sleep
Groups:
- Health Young Adults: Health Young adults, age 18-50 yrs
  hyperventilation and episodic hypoxia: noninvasive hyperventilation to determine apneic threshold; episodic hypoxia to determine long term facilitation
- Healthy Older Adults: Healthy Older adults, age >55-60yrs
  hyperventilation and episodic hypoxia: noninvasive hyperventilation to determine apneic threshold; episodic hypoxia to determine long term facilitation
- Total: Total of all reporting groups
Arm/Group | Health Young Adults | Healthy Older Adults | Total
Number analyzed (Participants) | 15 | 19 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (9.9) | 66.9 (5.4) | 48.3 (17.6)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Participants with data available were included in the analysis
  Participants
    Apneic Threshold & CO2 Reserve Analysis Population: number analyzed (Participants) | 15 | 10 | 25
    Apneic Threshold & CO2 Reserve Analysis Population: Female | 8 | 6 | 14
    Apneic Threshold & CO2 Reserve Analysis Population: Male | 7 | 4 | 11
    LTF and Minute Ventilation Analysis Population: number analyzed (Participants) | 15 | 14 | 29
    LTF and Minute Ventilation Analysis Population: Female | NA — Long-term Facilitation (LTF) of Ventilation, Minute Ventilation Was Measured in Older Adults Only | 8 | NA — Total not calculated because data are not available (NA) in one or more arms.
    LTF and Minute Ventilation Analysis Population: Male | NA — Long-term Facilitation (LTF) of Ventilation, Minute Ventilation Was Measured in Older Adults Only | 6 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Hypoxic Ventilatory Response Analysis Population: number analyzed (Participants) | 10 | 13 | 23
    Hypoxic Ventilatory Response Analysis Population: Female | 6 | 7 | 13
    Hypoxic Ventilatory Response Analysis Population: Male | 4 | 6 | 10
    Brief Hyperoxia Response Analysis Population: number analyzed (Participants) | 9 | 10 | 19
    Brief Hyperoxia Response Analysis Population: Female | 3 | 6 | 9
    Brief Hyperoxia Response Analysis Population: Male | 6 | 4 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 15 | 19 | 34
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 26.4 (2.4) | 27.3 (3.2) | 26.8 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Apneic Threshold (AT) and Carbon-dioxide (CO2) Reserve
Description: The AT was defined as the end-tidal (PETCO2) that demarcated the central apnea closest to the eupneic PETCO2. The CO2 reserve was defined as the difference in PETCO2 between eupnea and AT.
Time Frame: 4-6 wks for each participant
Population: Older adults : n=10, 6 females/4 males Young n=15, 8 females/ 7 males; participants with data available were included in the analysis
Measure: Mean (Standard Error); unit: mm Hg
Groups:
- Healthy Young Adults: Young adults, age 18-50 yrs
  hyperventilation and episodic hypoxia: noninvasive hyperventilation to determine apneic threshold; episodic hypoxia to determine long term facilitation
- Healthy Old Adults: Older adults, age >60 yrs
  hyperventilation and episodic hypoxia: noninvasive hyperventilation to determine apneic threshold; episodic hypoxia to determine long term facilitation
Arm/Group | Healthy Young Adults | Healthy Old Adults
Number analyzed (Participants) | 15 | 10
mm Hg
  Apneic Threshold | 39.8 (0.9) | 36.7 (1.3)
  Carbox-dioxide reserve | -4.1 (0.4) | -2.6 (0.4)
Statistical Analysis 1: Comparison: Healthy Young Adults vs Healthy Old Adults; T- test was conducted to compare the 2 groups; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Primary Outcome: Long-term Facilitation (LTF) of Ventilation, Minute Ventilation Was Measured in Older Adults Only
Description: Episodic hypoxia (EH) leads to sustained elevation of the ventilatory motor output, referred to as LTF, an excitatory mechanism characterized by a sustained elevation in ventilatory motor output following EH. Minute ventilation during recovery period after multiple trials of EH. This is reported in older adults on this grant.
Time Frame: 4-6 wks for each participant
Population: Older adults 8 women/6 men;participants with data available were included in the analysis
Measure: Mean (Standard Error); unit: percentage of control minute ventilation
Groups:
- Healthy Older Adults: Older adults
Arm/Group | Healthy Older Adults
Number analyzed (Participants) | 14
percentage of control minute ventilation | 94.4 (3.5)
Statistical Analysis 1: Comparison: Healthy Older Adults; Test type: Superiority or Other; p < 0.05, ANOVA; Compares control vs hypoxia trials vs recovery post-hypoxia

3. Secondary Outcome: Hypoxic Ventilatory Response
Description: Hypoxic ventilatory response was calculated as the change in minuted ventilation for a change in oxygen saturation during each hypoxia trial.
Time Frame: 4-6 wks for each participant
Population: older adults: 7 women/6 men; young adults: 6 women/4 men;participants with data available were included in the analysis
Measure: Mean (Standard Error); unit: Liter/minute/%saturation
Groups:
- Healthy Young Adults: Young adults
Arm/Group | Healthy Young Adults | Healthy Older Adults
Number analyzed (Participants) | 13 | 10
Liter/minute/%saturation | 0.21 (0.05) | 0.53 (0.36)
Statistical Analysis 1: Comparison: Healthy Young Adults vs Healthy Older Adults; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

4. Secondary Outcome: Brief Hyperoxia Response
Description: Brief hyperoxia response was the nadir minute ventilation achieved immediately upon exposure to brief hyperoxia expressed as a percent of eupneic minuted ventilation.
Time Frame: 4-6 wks for each participant
Population: young adults: 3 women/6 men; older adults: 6 women/4 men; participants with data available were included in the analysis
Measure: Mean (Standard Error); unit: percentage of eupneic minute ventilaion
Arm/Group | Healthy Young Adults | Healthy Older Adults
Number analyzed (Participants) | 9 | 10
percentage of eupneic minute ventilaion | 89.7 (8.4) | 79.6 (9.6)
Statistical Analysis 1: Comparison: Healthy Young Adults vs Healthy Older Adults; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: The participants were monitored throughout the study 2008 to 2013. Safety monitoring board also reviewed the study.
Groups:
- Healthy Older Adults: Older adults, age >55-60 years
  hyperventilation and episodic hypoxia: noninvasive hyperventilation to determine apneic threshold; episodic hypoxia to determine long term facilitation
Arm/Group | Healthy Young Adults | Healthy Older Adults
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/42
Other Adverse Events (participants affected / at risk) | 0/50 | 0/42

LIMITATIONS AND CAVEATS:
Participants who could not maintain stable sleep could not be included in the analyses. Participants also dropped out after the initial diagnostic sleep study as they did not want to continue the experimental arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes